CLINICAL TRIAL: NCT07148206
Title: Dronabinol and Epidiolex to Manage Uncontrolled Residual Symptoms of Buprenorphine Initiation Trial
Acronym: DEMURE
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2025-17060
Record Dates: First submitted 2025-08-21; First posted 2025-08-29 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Opioid Use Disorder
Keywords: Buprenorphine; delta-9-Tetrahydrocannabinol (THC); Cannabidiol (CBD); Cannabinoids; Opioid Use; Opioid Withdrawal; Retention to Treatment
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Dronabinol; Cannabidiol; Solutions

STUDY DESIGN:
Intervention Model Description: 1:1 randomization
Who Masked: Participant, Care Provider, Investigator
Masking Description: All products will be blinded to participants and research staff except for the study statistician and partnering pharmacists. Subject treatment assignments will remain blinded until the final subject has completed follow up and all data has been recorded and validated.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dronabinol + Epidiolex Arm (Experimental): Dronabinol (THC) will be dosed every 12 hours. To limit potential adverse effects, the dose of dronabinol will be titrated up gradually over 15 days to a final daily dose of 20 mg (10 mg every 12 hours). This final dosage will be administered twice daily from Day 16 to Week 8.
  Epidiolex (CBD) will also be dosed every 12 hours. To limit potential adverse effects, the dose of Epidiolex will be titrated up gradually over 15 days to a final dose of 400 mg every 12 hours. Participants will start off taking 200 mg daily (100 mg every 12 hours) for 5 days, then uptitrate to 400 mg (200 mg every 12 hours) for 5 days, then uptitrate to 600 mg for 5 days (300 mg every 12 hours), and finally 800 mg from day 16 through week 8 (400 mg every 12 hours).
  Interventions: Drug: Dronabinol Capsules; Drug: Epidiolex 100 mg/mL Oral Solution
- Placebo Arm (Placebo Comparator): Placebo Dronabinol capsules will be labeled and identical in appearance to dronabinol capsules. They will be made of pearl capsules filled with lactose by Montefiore's Investigational Drug Pharmacy team.
  Placebo Epidiolex oral solution will be made up of ethanol (79.0 mg/mL), sucralose (0.5 mg/mL), strawberry flavor (0.2 mg/mL), and refined sesame oil (to a volume of 1 mL). This mixture will be identical in appearance, taste, and composition of Epidiolex, except for the active ingredient of pure CBD.
  Interventions: Other: Placebo Dronabinol; Other: Placebo Epidiolex

INTERVENTIONS:
Drug: Dronabinol Capsules — Dronabinol is a synthetic form of THC. Dronabinol is eliminated in a biphasic manner, with an initial half-life of 25-36 hours.
  Other Names: Marinol
  Arms: Dronabinol + Epidiolex Arm
Drug: Epidiolex 100 mg/mL Oral Solution — Epidiolex is an oral solution (100 mg/mL) which rapidly appears in plasma, reaches peak plasma concentration in 3-4 hours and has a half-life of 18-32 hours.
  Other Names: Cannabidiol (CBD)
  Arms: Dronabinol + Epidiolex Arm
Other: Placebo Dronabinol — Placebo capsules
  Arms: Placebo Arm
Other: Placebo Epidiolex — Placebo oral solution
  Arms: Placebo Arm

SUMMARY:
The goal of this pilot study is to test novel, adjunctive pharmacotherapy for patients with opioid use disorder (POUD) who may be at risk for overdose and other poor opioid use disorder (OUD) outcomes even after initiating buprenorphine. The investigator team proposes to test the effectiveness of combined dronabinol (synthetic delta-9-tetrahydrocannabinol [THC]) and Epidiolex (cannabidiol [CBD]) - two FDA-approved cannabinoids - to improve retention in buprenorphine treatment and reduce opioid use among POUD who are early in treatment. POUD who are early in treatment are at a critical juncture-a moment of opportunity and motivation, but also of high risk of return to opioid use and loss to follow up.

DETAILED DESCRIPTION:
OUD and opioid overdose death rates remain shockingly high in the United States fueled by high potency opioids like fentanyl. Buprenorphine is an evidence-based therapy for OUD that reduces mortality, improves OUD outcomes, and is increasingly available. Three-month buprenorphine retention halves all-cause mortality; however, only 40-60% of POUD are retained in buprenorphine treatment for 3 or more months. Further, POUD who use fentanyl report protracted opioid withdrawal symptoms including anxiety, pain, insomnia, and opioid cravings, even months after reaching maximum doses of buprenorphine. Nearly 50% of POUD who use fentanyl return to use within 3 months.12 To improve success of buprenorphine treatment, new strategies for starting buprenorphine have emerged, such as low-dose initiation with ongoing opioid agonists, however, few interventions exist to improve treatment after starting buprenorphine, and those that exist are non-pharmacologic. Alpha-2-agonists (e.g., clonidine) reduce some withdrawal symptoms but can only be given for a short time without cardiac side effects. Pharmacologic adjuncts to buprenorphine are desperately needed to improve OUD outcomes in the fentanyl era.

Cannabis, the two key ingredients of which are THC and CBD, reduces opioid withdrawal in observational studies and thus has biologic plausibility for improving buprenorphine treatment retention. In two randomized trials, THC improved acute opioid withdrawal symptoms (e.g., muscle aches, muscle tension, and flu-like prodrome) a common driver of ongoing opioid use. THC is also effective in reducing acute and chronic pain in POUD another driver of ongoing use; however, patients receiving THC alone may experience adverse effects, such as panic, anxiety, and poor cognition. Co-administration with CBD may counteract these effects and maximize THC's benefits. In pre-clinical and clinical trials CBD reduces anxiety, pain, cue-induced opioid cravings, and attentional bias to drug-induced cues. When THC and CBD are co-administered, patients experience improved analgesic effects and reduced adverse effects. The overarching hypothesis of this study is that adjunctive dronabinol + Epidiolex improves buprenorphine retention and opioid use in POUD through reducing opioid withdrawal (including cravings, and pain).

The investigator team has developed an innovative 12-week pilot randomized trial of dronabinol + Epidiolex (versus placebo) as an adjunct to buprenorphine for OUD outcomes. 40 POUD participants within 21 days of buprenorphine initiation who are continuing either to use illicit opioids or to experience opioid withdrawal symptoms will be enrolled. Participants will be randomized to one of two arms as described in this registration. Study visits will occur at enrollment, and weeks 1, 2, 4, 8, and 12.

There are two overarching Aims in this study.

Aim 1: To determine the effectiveness and safety of 8- weeks of dronabinol + Epidiolex (vs. placebo) as an adjunct to buprenorphine in improving retention in OUD treatment and reducing opioid use. Hypothesis 1a: The dronabinol + Epidiolex (vs. placebo) group will have better 12-week retention in OUD treatment. Hypothesis 1b: The dronabinol + Epidiolex (vs. placebo) group will report less illicit opioid use. Hypothesis 2: The dronabinol + Epidiolex (vs. placebo) group will have no difference in significant adverse events or treatment limiting adverse events.

Aim 2: To explore the mechanism by which cannabinoids may improve OUD outcomes after buprenorphine initiation in POUD. The investigator team will explore how dronabinol + Epidiolex use are associated with change in opioid withdrawal symptoms, opioid cravings, and pain and whether these changes are associated with OUD outcomes. Hypothesis 3: The dronabinol + Epidiolex (vs. placebo) group will have fewer withdrawal symptoms, opioid cravings and pain, which will mediate the impact of cannabinoids on OUD outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Fluency in English and Spanish
* The Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) diagnosis of OUD
* Newly initiated on buprenorphine within 21 days
* Positive urine toxicology for opioids other than buprenorphine in the past week OR opioid withdrawal symptoms in the past week based on the Clinical Opioid Withdrawal Scale (COWS) >=5
* Any cannabis use in the past at or after the age of 18 years based on self-report

Exclusion Criteria:

* Urine toxicology positive for cannabinoids
* Inability to provide informed consent
* Liver tests (AST or ALT) >3 times the upper limit of normal, or a history of liver disease
* Pregnancy or breast/chest feeding
* Unstable cardiac disease, history of hypotension or syncope
* Psychotic disorder, or history of suicidal behavior and/or ideation
* Progressive neurological conditions, frequent falls, or history of epileptic seizures
* Severe alcohol use disorder, benzodiazepine use disorder or stimulant use disorder
* Other serious medical conditions that would be a contraindication to THC or CBD use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Retention in OUD Treatment | ~12 weeks following initiation of intervention
  Retention in OUD Treatment will be assessed as a dichotomous measure and will be based on the number of participants maintaining both an active buprenorphine prescription AND urine toxicology positive for buprenorphine at 12 weeks. The number/percentage of participants will be summarized by study arm.

SECONDARY OUTCOMES:
Retention in OUD Treatment | Baseline and ~1-week, 2-weeks, 4-weeks, and 8-weeks following initiation of intervention
  Retention in OUD Treatment will be assessed as a dichotomous measure and will be based on the number of participants maintaining both an active buprenorphine prescription AND urine toxicology positive for buprenorphine at 12 weeks. The number/percentage of participants will be summarized by study arm.
Opioid Use - Self Reported | Baseline and ~1-week, 2-weeks, 4-weeks, 8-weeks, and 12 weeks following initiation of intervention
  Self-reported opioid use will be assessed using the Timeline Follow-back (TLFB) calendar-based research tool. Using the TLFB methodology, participants will be provided with a calendar and asked to record, using a binary "Yes" or "No" response, whether opioid was used during each day over the prior 30-day period. Participants will be guided by a trained assessor during this process to help facilitate recall. If a participant's most recent study visit was within 30 days, then opioid use will be limited to the period of time since the last study visit. The number of days using opioids over the prior 30-day period will be summarized by study arm.
Opioid Use - Urine Toxicology | Baseline and ~2-weeks, 4-weeks, 8-weeks, and 12 weeks following initiation of intervention
  Opioid use will also be assessed using a urine toxicology immunoassay. Unobserved urine sample collection will be conducted at defined visits and samples will be analyzed to detect for the presence opioids and their metabolites. Results above the laboratory threshold for opiates will be reported as Either "Positive" or "Negative" and summarized by study arm at each timepoint.
Opioid Use Disorder Symptoms - Subjective Opiate Withdrawal Scale | Baseline and ~4-weeks, 8-weeks, and 12 weeks following initiation of intervention
  Opioid Use Disorder Symptoms will be assessed using the Subjective Opiate Withdrawal Scale (SOWS). The SOWS is a 16-item clinician administered scale designed to reproducibly rate the severity of opiate withdrawal symptoms. Participants rate each symptom on a 5-point scale ranging from 0 ("Not at all") to 4 ("Extremely") based on the intensity they are experiencing at the moment, yielding an overall possible range from 0-64, wherein higher scores are associated with more severe withdrawal symptoms. Specific scoring guideline categories include 1-10 = mild withdrawal; 11-20 = moderate withdrawal; 21-30+ = severe withdrawal. Mean scores will be summarized by study arm at each timepoint using basic descriptive statistics.
Opioid Use Disorder Symptoms - Opiate Craving Scale | Baseline and ~4-weeks, 8-weeks, and 12 weeks following initiation of intervention
  Opioid Use Disorder Symptoms will also be assessed using the 3-item Opiate Craving Scale. The Opiate Craving Scale is a clinician administered scale designed to evaluate opiate cravings over the prior week. Participants are asked to (1) "Please rate how strong your desire was to use in the past 24 hours." (2) "Please imagine yourself in the environment in which you previously used drugs or alcohol. If you were in this environment today, what is the likelihood you would use?" and (3) "Please rate how strong your urges are for drugs or alcohol when something in the environment reminds you of it." Each item is rated on a scale ranging from 0 to 9 and an average score from the 3 items is calculated. Higher scores are indicative of greater craving. Mean scores will be summarized by study arm using basic descriptive statistics.
Pain Severity | Baseline and ~1-week, 2-weeks, 4-weeks, 8-weeks, and 12 weeks following initiation of intervention
  Pain Severity will be assessed by administration of the Pain Severity questions within the Brief Pain Inventory-Short Form (BPI-SF). Pain severity over the prior 24 hours is calculated by averaging the ratings for worst, least, and average pain for the past week as well as current pain (four individual items on the BPI-SF). This results in a Pain Severity score ranging from 0-10, with higher scores being indicative of more severe pain. A score of 0 means "No pain" and a score of 10 means "Pain as bad as you can imagine." Scores will be summarized by study arm at each timepoint using basic descriptive statistics.
Pain Interference | Baseline and ~1-week, 2-weeks, 4-weeks, 8-weeks, and 12 weeks following initiation of intervention
  Pain Interference will be assessed using the corresponding Pain Interference questions within the Brief Pain Inventory-Short Form (BPI-SF). Pain interference over the prior 24 hours is calculated by averaging the ratings of the corresponding 7 items on the questionnaire to determine how much pain interferes with general activity, mood, walking, work, relations, sleep, and enjoyment of life. This results in a Pain Interference score ranging from 0-10, with higher scores indicating that the pain is more significantly interfering with daily activities. A score of 0 means "No Interference" and a score of 10 means "Pain completely interferes with daily activities." Scores will be summarized by study arm at each timepoint using basic descriptive statistics.
Panic Symptoms | Baseline and ~1-week, 2-weeks, 4-weeks, 8-weeks, and 12 weeks following initiation of intervention
  Panic symptoms will be assessed by administration of the Panic Disorder Severity Scale (PDSS). The PDSS is a seven-item self-report scale that measures the severity of panic attacks and panic disorder symptoms. Each of the 7 items is rated on a 5-point Likert scale ranging from 0 ("No/None/Not at all") to 4 ("Extreme/Extremely/Nearly constantly") yielding an overall possible scoring range of 0-28, such that higher scores are indicative of greater severity of panic disorder. Scores will be summarized by study arm at each timepoint using basic descriptive statistics.
Anxiety Symptoms | Baseline and ~4-weeks, 8-weeks, and 12 weeks following initiation of intervention
  Anxiety will be assessed by administration of the Generalized Anxiety Disorder 7-item (GAD-7) questionnaire. The GAD-7 is a seven-item screening tool used to assess the severity of generalized anxiety disorder over the prior two-week period. Each item on the questionnaire is rated on a 4-point Likert scale ranging from 0 ("Not at all") to 3 ("Nearly every day") yielding an overall possible scoring range of 0-21, such that higher scores are indicative of greater anxiety. Scores will be summarized by study arm at each timepoint using basic descriptive statistics.
Cognitive Function | Baseline and ~1-week, 2-weeks, 4-weeks, 8-weeks, and 12 weeks following initiation of intervention
  Cognitive Function will be assessed by administration of the Patient-Reported Outcomes Measurement Information System Cognitive Function (PROMIS-CF) questionnaire. The PROMIS-CF questionnaire is a 4-item patient-reported outcome measures that assesses self-perceived cognitive abilities in the domains of memory (2 items) and concentration (2 items). Responses are scored on a 5-point Likert scale ranging from 1-5, yielding a scoring range of 4-20. Using item-level calibrations, raw scores are then converted to T-scores. T-scores are standardized to a metric with a mean of 50 and a standard deviation of 10 for reference to a population. Higher scores on the PROMIS-CF indicate better perceived cognitive function. Scores will be summarized by study arm at each timepoint using basic descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Deepika Slawek, MD, MPH, MS, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Health System (Montefiore) Buprenorphine Treatment Network, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual Participant Data (IPD) Sharing Statement will be completed upon receipt of Notice of Award.

REFERENCES:
- [Background] The ASAM National Practice Guideline for the Treatment of Opioid Use Disorder: 2020 Focused Update. J Addict Med. 2020 Mar/Apr;14(2S Suppl 1):1-91. doi: 10.1097/ADM.0000000000000633. No abstract available. PMID 32511106
- [Background] Schwartz RP, Gryczynski J, O'Grady KE, Sharfstein JM, Warren G, Olsen Y, Mitchell SG, Jaffe JH. Opioid agonist treatments and heroin overdose deaths in Baltimore, Maryland, 1995-2009. Am J Public Health. 2013 May;103(5):917-22. doi: 10.2105/AJPH.2012.301049. Epub 2013 Mar 14. PMID 23488511
- [Background] Samples H, Williams AR, Crystal S, Olfson M. Impact Of Long-Term Buprenorphine Treatment On Adverse Health Care Outcomes In Medicaid. Health Aff (Millwood). 2020 May;39(5):747-755. doi: 10.1377/hlthaff.2019.01085. PMID 32364847
- [Background] Krawczyk N, Mojtabai R, Stuart EA, Fingerhood M, Agus D, Lyons BC, Weiner JP, Saloner B. Opioid agonist treatment and fatal overdose risk in a state-wide US population receiving opioid use disorder services. Addiction. 2020 Sep;115(9):1683-1694. doi: 10.1111/add.14991. Epub 2020 Feb 24. PMID 32096302
- [Background] Nunes EV, Comer SD, Lofwall MR, Walsh SL, Peterson S, Tiberg F, Hjelmstrom P, Budilovsky-Kelley NR. Extended-Release Injection vs Sublingual Buprenorphine for Opioid Use Disorder With Fentanyl Use: A Post Hoc Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2024 Jun 3;7(6):e2417377. doi: 10.1001/jamanetworkopen.2024.17377. PMID 38916892
- [Background] Mariani JJ, Dobbins RL, Heath A, Gray F, Hassman H. Open-label investigation of rapid initiation of extended-release buprenorphine in patients using fentanyl and fentanyl analogs. Am J Addict. 2024 Jan;33(1):8-14. doi: 10.1111/ajad.13484. Epub 2023 Nov 8. PMID 37936553
- [Background] Santo T Jr, Clark B, Hickman M, Grebely J, Campbell G, Sordo L, Chen A, Tran LT, Bharat C, Padmanathan P, Cousins G, Dupouy J, Kelty E, Muga R, Nosyk B, Min J, Pavarin R, Farrell M, Degenhardt L. Association of Opioid Agonist Treatment With All-Cause Mortality and Specific Causes of Death Among People With Opioid Dependence: A Systematic Review and Meta-analysis. JAMA Psychiatry. 2021 Sep 1;78(9):979-993. doi: 10.1001/jamapsychiatry.2021.0976. PMID 34076676
- [Background] Wyse JJ, Eckhardt A, Waller D, Gordon AJ, Shull S, Lovejoy TI, Mackey K, Morasco BJ. Patients' Perspectives on Discontinuing Buprenorphine for the Treatment of Opioid Use Disorder. J Addict Med. 2024 May-Jun 01;18(3):300-305. doi: 10.1097/ADM.0000000000001292. Epub 2024 Mar 18. PMID 38498620
- [Background] Reddon H, Lake S, Socias ME, Hayashi K, DeBeck K, Walsh Z, Milloy MJ. Cannabis use to manage opioid cravings among people who use unregulated opioids during a drug toxicity crisis. Int J Drug Policy. 2023 Sep;119:104113. doi: 10.1016/j.drugpo.2023.104113. Epub 2023 Jul 21. PMID 37481875
- [Background] Spadaro A, Sarker A, Hogg-Bremer W, Love JS, O'Donnell N, Nelson LS, Perrone J. Reddit discussions about buprenorphine associated precipitated withdrawal in the era of fentanyl. Clin Toxicol (Phila). 2022 Jun;60(6):694-701. doi: 10.1080/15563650.2022.2032730. Epub 2022 Feb 4. PMID 35119337
- [Background] Wakeman SE, Chang Y, Regan S, Yu L, Flood J, Metlay J, Rigotti N. Impact of Fentanyl Use on Buprenorphine Treatment Retention and Opioid Abstinence. J Addict Med. 2019 Jul/Aug;13(4):253-257. doi: 10.1097/ADM.0000000000000486. PMID 30550392
- [Background] Randhawa PA, Brar R, Nolan S. Buprenorphine-naloxone "microdosing": an alternative induction approach for the treatment of opioid use disorder in the wake of North America's increasingly potent illicit drug market. CMAJ. 2020 Jan 20;192(3):E73. doi: 10.1503/cmaj.74018. No abstract available. PMID 31959660
- [Background] Klaire S, Zivanovic R, Barbic SP, Sandhu R, Mathew N, Azar P. Rapid micro-induction of buprenorphine/naloxone for opioid use disorder in an inpatient setting: A case series. Am J Addict. 2019 Jul;28(4):262-265. doi: 10.1111/ajad.12869. Epub 2019 Mar 22. PMID 30901127
- [Background] Azar P, Schneiderman H, Barron H, Wong JSH, Meyer M, Newman-Azar D, Narimani M, Ignaszewski MJ, Mathew N, Mullen R, Krausz RM, Maharaj AR. Rapid induction of transdermal buprenorphine to subcutaneous extended-release buprenorphine for the treatment of opioid use disorder. Addict Sci Clin Pract. 2024 Jun 18;19(1):50. doi: 10.1186/s13722-024-00479-1. PMID 38886826
- [Background] D'Onofrio G, Perrone J, Hawk KF, Cowan E, McCormack R, Coupet E Jr, Owens PH, Martel SH, Huntley K, Walsh SL, Lofwall MR, Herring A; ED-INNOVATION Investigators. Early emergency department experience with 7-day extended-release injectable buprenorphine for opioid use disorder. Acad Emerg Med. 2023 Dec;30(12):1264-1271. doi: 10.1111/acem.14782. Epub 2023 Aug 22. PMID 37501652
- [Background] Rosic T, Kapoor R, Panesar B, Naji L, Chai DB, Sanger N, Marsh DC, Worster A, Thabane L, Samaan Z. The association between cannabis use and outcome in pharmacological treatment for opioid use disorder. Harm Reduct J. 2021 Feb 23;18(1):24. doi: 10.1186/s12954-021-00468-6. PMID 33622351
- [Background] Lucas P, Walsh Z. Medical cannabis access, use, and substitution for prescription opioids and other substances: A survey of authorized medical cannabis patients. Int J Drug Policy. 2017 Apr;42:30-35. doi: 10.1016/j.drugpo.2017.01.011. Epub 2017 Feb 9. PMID 28189912
- [Background] Bergeria CL, Huhn AS, Dunn KE. The impact of naturalistic cannabis use on self-reported opioid withdrawal. J Subst Abuse Treat. 2020 Jun;113:108005. doi: 10.1016/j.jsat.2020.108005. Epub 2020 Mar 30. PMID 32359667
- [Background] Bisaga A, Sullivan MA, Glass A, Mishlen K, Pavlicova M, Haney M, Raby WN, Levin FR, Carpenter KM, Mariani JJ, Nunes EV. The effects of dronabinol during detoxification and the initiation of treatment with extended release naltrexone. Drug Alcohol Depend. 2015 Sep 1;154:38-45. doi: 10.1016/j.drugalcdep.2015.05.013. Epub 2015 Jul 8. PMID 26187456
- [Background] Lofwall MR, Babalonis S, Nuzzo PA, Elayi SC, Walsh SL. Opioid withdrawal suppression efficacy of oral dronabinol in opioid dependent humans. Drug Alcohol Depend. 2016 Jul 1;164:143-150. doi: 10.1016/j.drugalcdep.2016.05.002. Epub 2016 May 10. PMID 27234658
- [Background] Whiting PF, Wolff RF, Deshpande S, Di Nisio M, Duffy S, Hernandez AV, Keurentjes JC, Lang S, Misso K, Ryder S, Schmidlkofer S, Westwood M, Kleijnen J. Cannabinoids for Medical Use: A Systematic Review and Meta-analysis. JAMA. 2015 Jun 23-30;313(24):2456-73. doi: 10.1001/jama.2015.6358. PMID 26103030
- [Background] National Academies of Sciences, Engineering, and Medicine; Health and Medicine Division; Board on Population Health and Public Health Practice; Committee on the Health Effects of Marijuana: An Evidence Review and Research Agenda. The Health Effects of Cannabis and Cannabinoids: The Current State of Evidence and Recommendations for Research. Washington (DC): National Academies Press (US); 2017 Jan 12. Available from http://www.ncbi.nlm.nih.gov/books/NBK423845/ PMID 28182367
- [Background] McDonagh MS, Morasco BJ, Wagner J, Ahmed AY, Fu R, Kansagara D, Chou R. Cannabis-Based Products for Chronic Pain : A Systematic Review. Ann Intern Med. 2022 Aug;175(8):1143-1153. doi: 10.7326/M21-4520. Epub 2022 Jun 7. PMID 35667066
- [Background] Dennis BB, Bawor M, Naji L, Chan CK, Varenbut J, Paul J, Varenbut M, Daiter J, Plater C, Pare G, Marsh DC, Worster A, Desai D, Thabane L, Samaan Z. Impact of Chronic Pain on Treatment Prognosis for Patients with Opioid Use Disorder: A Systematic Review and Meta-analysis. Subst Abuse. 2015 Sep 10;9:59-80. doi: 10.4137/SART.S30120. eCollection 2015. PMID 26417202
- [Background] Le K, Le KDR, Nguyen J, Hua J, Munday S. The Role of Medicinal Cannabis as an Emerging Therapy for Opioid Use Disorder. Pain Ther. 2024 Jun;13(3):435-455. doi: 10.1007/s40122-024-00599-1. Epub 2024 Apr 27. PMID 38676910
- [Background] Hurd YL, Spriggs S, Alishayev J, Winkel G, Gurgov K, Kudrich C, Oprescu AM, Salsitz E. Cannabidiol for the Reduction of Cue-Induced Craving and Anxiety in Drug-Abstinent Individuals With Heroin Use Disorder: A Double-Blind Randomized Placebo-Controlled Trial. Am J Psychiatry. 2019 Nov 1;176(11):911-922. doi: 10.1176/appi.ajp.2019.18101191. Epub 2019 May 21. PMID 31109198
- [Background] Suzuki J, Prostko S, Szpak V, Chai PR, Spagnolo PA, Tenenbaum RE, Ahmed S, Weiss RD. Impact of cannabidiol on reward- and stress-related neurocognitive processes among individuals with opioid use disorder: A pilot, double-blind, placebo-controlled, randomized cross-over trial. Front Psychiatry. 2023 Mar 30;14:1155984. doi: 10.3389/fpsyt.2023.1155984. eCollection 2023. PMID 37065899
- [Background] Cunningham CO, Starrels JL, Zhang C, Bachhuber MA, Sohler NL, Levin FR, Minami H, Slawek DE, Arnsten JH. Medical Marijuana and Opioids (MEMO) Study: protocol of a longitudinal cohort study to examine if medical cannabis reduces opioid use among adults with chronic pain. BMJ Open. 2020 Dec 29;10(12):e043400. doi: 10.1136/bmjopen-2020-043400. PMID 33376181
- [Background] McKnight C, Weng CA, Reynoso M, Kimball S, Thompson LM, Jarlais DD. Understanding intentionality of fentanyl use and drug overdose risk: Findings from a mixed methods study of people who inject drugs in New York City. Int J Drug Policy. 2023 Aug;118:104063. doi: 10.1016/j.drugpo.2023.104063. Epub 2023 Jun 2. PMID 37270373
- [Background] National Academies of Sciences, Engineering, and Medicine; Health and Medicine Division; Board on Health Sciences Policy; Committee on Medication-Assisted Treatment for Opioid Use Disorder; Mancher M, Leshner AI, editors. Medications for Opioid Use Disorder Save Lives. Washington (DC): National Academies Press (US); 2019 Mar 30. Available from http://www.ncbi.nlm.nih.gov/books/NBK538936/ PMID 30896911
- [Background] MacArthur GJ, Minozzi S, Martin N, Vickerman P, Deren S, Bruneau J, Degenhardt L, Hickman M. Opiate substitution treatment and HIV transmission in people who inject drugs: systematic review and meta-analysis. BMJ. 2012 Oct 3;345:e5945. doi: 10.1136/bmj.e5945. PMID 23038795
- [Background] De Maeyer J, Vanderplasschen W, Broekaert E. Quality of life among opiate-dependent individuals: A review of the literature. Int J Drug Policy. 2010 Sep;21(5):364-80. doi: 10.1016/j.drugpo.2010.01.010. Epub 2010 Feb 20. PMID 20172706
- [Background] Platt L, Minozzi S, Reed J, Vickerman P, Hagan H, French C, Jordan A, Degenhardt L, Hope V, Hutchinson S, Maher L, Palmateer N, Taylor A, Bruneau J, Hickman M. Needle syringe programmes and opioid substitution therapy for preventing hepatitis C transmission in people who inject drugs. Cochrane Database Syst Rev. 2017 Sep 18;9(9):CD012021. doi: 10.1002/14651858.CD012021.pub2. PMID 28922449
- [Background] Coe MA, Lofwall MR, Walsh SL. Buprenorphine Pharmacology Review: Update on Transmucosal and Long-acting Formulations. J Addict Med. 2019 Mar/Apr;13(2):93-103. doi: 10.1097/ADM.0000000000000457. PMID 30531584
- [Background] Volpe DA, McMahon Tobin GA, Mellon RD, Katki AG, Parker RJ, Colatsky T, Kropp TJ, Verbois SL. Uniform assessment and ranking of opioid mu receptor binding constants for selected opioid drugs. Regul Toxicol Pharmacol. 2011 Apr;59(3):385-90. doi: 10.1016/j.yrtph.2010.12.007. Epub 2011 Jan 6. PMID 21215785
- [Background] Samuels EA, Martin AF. Beyond the Waiver: Multilevel Interventions Needed to Expand Buprenorphine Treatment. JAMA Netw Open. 2022 May 2;5(5):e2212425. doi: 10.1001/jamanetworkopen.2022.12425. No abstract available. PMID 35552731
- [Background] Biondi BE, Vander Wyk B, Schlossberg EF, Shaw A, Springer SA. Factors associated with retention on medications for opioid use disorder among a cohort of adults seeking treatment in the community. Addict Sci Clin Pract. 2022 Mar 7;17(1):15. doi: 10.1186/s13722-022-00299-1. PMID 35255967
- [Background] Simpson SA, Hordes M, Blum J, Rinehart D, Al-Tayyib A. Barriers to Engagement in Opioid Use Disorder Treatment After Buprenorphine Induction. J Addict Med. 2022 Jul-Aug 01;16(4):479-482. doi: 10.1097/ADM.0000000000000943. Epub 2021 Dec 23. PMID 34954744
- [Background] O'Connor AM, Cousins G, Durand L, Barry J, Boland F. Retention of patients in opioid substitution treatment: A systematic review. PLoS One. 2020 May 14;15(5):e0232086. doi: 10.1371/journal.pone.0232086. eCollection 2020. PMID 32407321
- [Background] Stein MD, VanNoppen D, Herman DS, Anderson BJ, Conti M, Bailey GL. Retention in care for persons with opioid use disorder transitioning from sublingual to injectable buprenorphine. J Subst Abuse Treat. 2022 May;136:108661. doi: 10.1016/j.jsat.2021.108661. Epub 2021 Nov 14. PMID 34801283
- [Background] Ricarte A, Dalton JAR, Giraldo J. Structural Assessment of Agonist Efficacy in the mu-Opioid Receptor: Morphine and Fentanyl Elicit Different Activation Patterns. J Chem Inf Model. 2021 Mar 22;61(3):1251-1274. doi: 10.1021/acs.jcim.0c00890. Epub 2021 Jan 15. PMID 33448226
- [Background] Armenian P, Vo KT, Barr-Walker J, Lynch KL. Fentanyl, fentanyl analogs and novel synthetic opioids: A comprehensive review. Neuropharmacology. 2018 May 15;134(Pt A):121-132. doi: 10.1016/j.neuropharm.2017.10.016. Epub 2017 Oct 14. PMID 29042317
- [Background] Chambers LC, Hallowell BD, Zullo AR, Paiva TJ, Berk J, Gaither R, Hampson AJ, Beaudoin FL, Wightman RS. Buprenorphine Dose and Time to Discontinuation Among Patients With Opioid Use Disorder in the Era of Fentanyl. JAMA Netw Open. 2023 Sep 5;6(9):e2334540. doi: 10.1001/jamanetworkopen.2023.34540. PMID 37721749
- [Background] Northrup TF, Stotts AL, Green C, Potter JS, Marino EN, Walker R, Weiss RD, Trivedi M. Opioid withdrawal, craving, and use during and after outpatient buprenorphine stabilization and taper: a discrete survival and growth mixture model. Addict Behav. 2015 Feb;41:20-8. doi: 10.1016/j.addbeh.2014.09.021. Epub 2014 Sep 28. PMID 25282598
- [Background] Luba R, Jones J, Choi CJ, Comer S. Fentanyl withdrawal: Understanding symptom severity and exploring the role of body mass index on withdrawal symptoms and clearance. Addiction. 2023 Apr;118(4):719-726. doi: 10.1111/add.16100. Epub 2022 Dec 13. PMID 36444486
- [Background] Bolshakova M, Simpson KA, Ganesh SS, Goldshear JL, Page CJ, Bluthenthal RN. The fentanyl made me feel like I needed more methadone": changes in the role and use of medication for opioid use disorder (MOUD) due to fentanyl. Harm Reduct J. 2024 Aug 24;21(1):156. doi: 10.1186/s12954-024-01075-x. PMID 39182110
- See also: Arnsten JH. Does Medical Cannabis Reduce Opioid Use in Adults With Pain — https://www.clinicaltrials.gov/study/NCT04308148
- See also: Slawek DE. Pain, Inflammation, and Cannabis in HIV — https://classic.clinicaltrials.gov/ct2/show/NCT05554146
- See also: Withdrawal Management. In: Clinical Guidelines for Withdrawal Management and Treatment of Drug Dependence in Closed Settings. World Health Organization; 2009. — https://www.ncbi.nlm.nih.gov/books/NBK310652/